CLINICAL TRIAL: NCT06723678
Title: Radiographic Evaluation of Crestal Bone Changes Around Implants in Patients Treated With Delayed Loaded All on Four (Randomized Clinical Trail)
Brief Title: Evaluation of Bone Changes Around Implants in Patients Treated With All on Four
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Noha Taha Kamel Taha Alloush, Lecturer, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-PD-24-28
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Edentulous Alveolar Ridge In Mandible; Complete Edentulism; All on Four Technique; Dental Implant; Edentulous Jaws; Edentulous Mouth
Keywords: Completely edentulous patients; Dental Implants; All on four technique; Fixed Detachable Prosthesis; screw retained prosthesis
MeSH Terms: conditions — Jaw, Edentulous; Mouth, Edentulous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two distally inclined 45-degree angle posterior implants. (Experimental): During the surgery, two axially placed anterior implants and two distally inclined 45-degree angle posterior implants.
  Interventions: Procedure: Two distally inclined 45-degree angle posterior implants
- Two distally inclined 30-degree angle posterior implants. (Active Comparator): During the surgery, two axially placed anterior implants and two distally inclined 30-degree angle posterior implants.
  Interventions: Procedure: Two distally inclined 30-degree angle posterior implants

INTERVENTIONS:
Procedure: Two distally inclined 45-degree angle posterior implants — During the surgery, two axially placed anterior implants and two distally inclined 45-degree angle posterior implants will be placed, after healing period, All on-4 screw-retained prosthesis will be delivered to the patients.
  Arms: Two distally inclined 45-degree angle posterior implants.
Procedure: Two distally inclined 30-degree angle posterior implants — During the surgery, two axially placed anterior implants and two distally inclined 30-degree angle posterior implants will be placed, after healing period, All on-4 screw-retained prosthesis will be delivered to the patients
  Arms: Two distally inclined 30-degree angle posterior implants.

SUMMARY:
The Goal of the clinical trail is to evaluate the Bone height changes around two axially placed anterior implants and two distally inclined 30-degree angle posterior implants in comparison to two axially placed anterior implants and two distally inclined 45-degree angle posterior implants using cone beam CT (CBCT).

Patients will visit the clinic after the surgery and after the framework and denture insertion for check ups and during the follow up periods ( at denture insertion, 6 months and 12 months)

DETAILED DESCRIPTION:
All patients will receive upper complete dentures and mandibular All on-4 screw-retained prosthesis. The upper complete denture will be mucosa supported and the lower will be All on-4 screw-retained prosthesis. Patients will be divided into two equal groups; Group I will receive two axially placed anterior implants and two distally inclined 30-degree angle posterior implants, while Group II will receive two axially placed anterior implants and two distally inclined 45-degree angle posterior implants.

Both groups will be functionally loaded after three months of insertion. Bone height changes around axial and distally inclined implants will be evaluated using cone beam CT (CBCT), All records will be taken at time of denture insertion, 6 and 12 months later.

ELIGIBILITY:
Inclusion Criteria:

* All patients' ages must range from 50-65 years old.
* All patients' ridges should be covered with firm mucosa free from any signs of inflammation or ulceration and exhibit adequate height and width of the residual alveolar ridge.
* Patients should be free from any metabolic or bone disorders that contraindicate implant installation.
* All patients must have sufficient inter arch space

Exclusion Criteria:

* Patients with oral or systemic diseases.
* Patients with xerostomia or excessive salivation.
* Patients with parafunctional habits (bruxism or clenching).
* Heavy smoker or alcoholic patients.
* Patients with history of temporo-mandibular dysfunction.
* Patients with brain disorders or psychiatric disorders

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Bone Height Changes | All records will be taken at time of denture insertion, 6 and 12 months later.
  Bone height changes around axially placed anterior implants and distally inclined posterior implants will be evaluated using cone beam CT (CBCT)

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University Girls Branch, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Clinical Study Report
Supporting Information: Study Protocol, CSR
Time Frame: Start Date: After publication End Date: 10 years
Access Criteria: After publication through the corresponding author